CLINICAL TRIAL: NCT03544814
Title: EGFR Tyrosine Kinase Inhibitor Combined With Concurrent or Sequential Chemotherapy for Advanced Lung Cancer Patients of Gradual Progression After First-line EGFR-TKI Therapy: a Randomized Controlled Study
Brief Title: EGFR-TKI Combined With Concurrent or Sequential Chemotherapy for Patients of Gradual Progression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Tianqing Chu, Associate Chief Physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chest006
Record Dates: First submitted 2018-05-21; First posted 2018-06-04 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2015-01

CONDITIONS: Lung Adenocarcinoma; EGFR Activating Mutation
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Pemetrexed; Cisplatin; Drug Therapy

ARMS (2):
- Concurrent therapy group (Experimental): Icotinib combined with pemetrexed plus cisplatin.
  Interventions: Drug: icotinib combined with pemetrexed plus cisplatin
- Sequential therapy group (Experimental): First icotinib and then pemetrexed plus cisplatin.
  Interventions: Drug: first icotinib and then pemetrexed plus cisplatin

INTERVENTIONS:
Drug: icotinib combined with pemetrexed plus cisplatin — Continued using the icotinib (125 mg/time, 3 times/day every day) combined with Pemetrexed (500 mg/㎡ on day 1) plus cisplatin (75mg/m2 on day 1) and repeat every four weeks for up to six cycles and then continue to receive pemetrexed combined with icotinib every four weeks.
  Other Names: EGFR-TKI combined with chemotherapy
  Arms: Concurrent therapy group
Drug: first icotinib and then pemetrexed plus cisplatin — Continued using the icotinib (125 mg/time, 3 times/day every day)) alone until the investigator judged that continuation was adiaphorous, and switched to Pemetrexed (500 mg/㎡ on day 1) plus cisplatin (75mg/m2 on day 1) alone, repeat every four weeks for up to six cycles and then continue to receive pemetrexed every four weeks.
  Other Names: chemotherapy
  Arms: Sequential therapy group

SUMMARY:
To compare the efficacy of simultaneous EGFR-TKI and chemotherapy with that of sequential treatment after patients gradually progressed from first-line EGFR-TKI treatment.

Patients who had gradual progression and EGFR-T790M mutation-negative were randomly divided into two groups: in concurrent group, patients were treated with pemetrexed plus cisplatin along with the same EGFR-TKI; in sequential group, patients continued with EGFR-TKI until the disease progressed again according to the RECIST criteria, and then switched to chemotherapy. We evaluated progression-free survival (PFS) and overall survival (OS) time of patients. For sequential group, PFS was PFS1 (gradual progression to discontinue EGFR-TKI) plus PFS2 (chemotherapy alone).

DETAILED DESCRIPTION:
According to previous reports, when non-small cell lung cancer (NSCLC) patients with EGFR mutations gradually progressed after initial EGFR tyrosine-kinase inhibitor (TKI) treatment, continuing TKI therapy may be beneficial. We aimed to compare the efficacy of simultaneous EGFR-TKI and chemotherapy with that of sequential treatment after patients gradually progressed from first-line EGFR-TKI treatment.

Patients who had gradual progression and EGFR-T790M mutation-negative were randomly divided into two groups: in concurrent group, patients were treated with pemetrexed plus cisplatin along with the same EGFR-TKI; in sequential group, patients continued with EGFR-TKI until the disease progressed again according to the RECIST criteria, and then switched to chemotherapy. We evaluated progression-free survival (PFS) and overall survival (OS) time of patients. For sequential group, PFS was PFS1 (gradual progression to discontinue EGFR-TKI) plus PFS2 (chemotherapy alone). Objective response rate (ORR), disease control rate (DCR), overall survival (OS), and safety were also evaluated.

ELIGIBILITY:
Inclusion criteria：

1. Patients had to voluntarily join the study and give written informed consent for the study
2. Histologically documented, unresectable, inoperable, locally advanced, recurrent or metastatic stage IIIB or IV adenocarcinoma.
3. A cytologic diagnosis is acceptable (i.e., FNA or pleural fluid cytology)
4. Sensitive EGFR mutations (exon 19 deletion or L858R mutation in exon 21)
5. At least one measurable lesion meeting Response Evaluation Criteria in Solid Tumours (RECIST) criteria.
6. Patients achieved the gradual progression after first-line EGFR-TKI therapy.

The criteria of gradual progression:

1. disease control≥6 months with EGFR-TKI treatment;
2. compared with the previous assessment，no significant increment of tumor burden and progressive involvement of non-target lesions with a score ≤2;
3. symptom scored≤1. 7) Patients did not achieve acquired EGFR-T790M mutation assessed by ARMS, next-generation sequencing (NGS) or droplet digital PCR (ddPCR) after first-line EGFR-TKI therapy 8) Patients did not receive any chemotherapy previously 9) Able to comply with study and follow-up procedures 10) Age >=18 years, ECOG PS: 0~2, estimated survival duration more than 3 months； 11) Major organ function

Exclusion criteria：

1. Other types of non-small cell lung cancer except adenocarcinoma and Small cell lung cancer（including patients with mixed small cell lung cancer and non-small cell lung cancer）；
2. Evidence of other types of non-small cell lung cancer except adenocarcinoma, small cell, carcinoid, or mixed small cell/non-small cell histology
3. EGFR wild-type patients, or patients with rare EGFR mutations or complex EGFR mutations
4. Patients achieved the dramatic progression after first-line EGFR-TKI therapy. The criteria of dramatic progression
5. Patients achieved the local progression after first-line EGFR-TKI therapy. The criteria of local progression
6. Patients achieved acquired EGFR-T790M mutation assessed by ARMS, next-generation sequencing (NGS) or droplet digital PCR (ddPCR) after first-line EGFR-TKI therapy
7. Previously (within 5 years) or presently suffering from other malignancies
8. A in situ，non-melanoma skin cancers and superficial bladder cancer
9. Unstable systemic disease
10. History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications
11. Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, or prior surgical procedures affecting absorption
12. Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 16 months
  Radiographic assessments were performed when enrolled and every 8 weeks until disease progression after chemotherapy according to RECIST version 1.1. After PD, collect the survival information every 16 weeks until death or withdrawal of study consent.

SECONDARY OUTCOMES:
overall survival (OS) | 32 months
  Radiographic assessments were performed when enrolled and every 8 weeks until disease progression after chemotherapy according to RECIST version 1.1. After PD, collect the survival information every 16 weeks until death or withdrawal of study consent.

CONTACTS AND LOCATIONS:
Overall Officials: Tianqing Chu, Principal Investigator — Shanghai Chest Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang JJ, Chen HJ, Yan HH, Zhang XC, Zhou Q, Su J, Wang Z, Xu CR, Huang YS, Wang BC, Yang XN, Zhong WZ, Nie Q, Liao RQ, Jiang BY, Dong S, Wu YL. Clinical modes of EGFR tyrosine kinase inhibitor failure and subsequent management in advanced non-small cell lung cancer. Lung Cancer. 2013 Jan;79(1):33-9. doi: 10.1016/j.lungcan.2012.09.016. Epub 2012 Oct 15. PMID 23079155

DOCUMENTS (2):
  • Informed Consent Form (2015-04-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03544814/ICF_000.pdf
  • Study Protocol (2015-04-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03544814/Prot_001.pdf